CLINICAL TRIAL: NCT02254434
Title: An Open-label Single-dose Pharmacokinetic Study of an Oral Formulation in Tablets Containing Eltrombopag 50 mg (Revolade, Glaxosmithkline Mexico, S.A. De C.V.) in Healthy Volunteers Under Fasting Conditions
Brief Title: A Pharmacokinetic Study of Eltrombopag 50 Milligram (mg) in Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200338
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cirrhosis, Liver
Keywords: eltrombopag 50 mg; healthy volunteers; pharmacokinetic; single-dose; Open-label; fasting
MeSH Terms: conditions — Liver Cirrhosis; Fasting | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eltrombopag 50 mg (Experimental): Each volunteer will receive orally, single dose of tablet eltrombopag 50 mg under fasting conditions
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag 50 mg per tablet for oral route of administration will be sourced locally

SUMMARY:
This study evaluates pharmacokinetics of eltrombopag 50 mg after the oral administration in Mexican healthy volunteers under fasting conditions. The study will be an open label, single dose study with 26 subjects planned to be enrolled. Healthy subjects (male and female) aged between 18 - 50 years of age (inclusive) and a Body Mass Index within the range of 18-27.0 kg/meter (m)^2 (inclusive) were enrolled according to Quetelet. REVOLADE is a registered trademark of the GSK group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' participation must be voluntary according to the General Health Law and an informed consent form must be obtained for each subject before their participation. Compliance to Helsinki´s Declaration, its Japan Review and good clinical practice (GCP) should be followed.
* Mexican male and female healthy volunteers with 18 to 50 years old will be included. A female subject is eligible to participate if she is of, Non-childbearing potential defined as pre menopausal females with a documented tubal ligation or hysterectomy (for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] > 40 milliinternational units per milliliter (MlU/ml) and estradiol < 40 picogram per milliliter [pg/ml] [<147 picomole per liter (pmol/L)] is confirmatory). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods as described by the Investigator/designee, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method). Child-bearing potential with negative pregnancy test as determined by (serum or urine) human chorionic gonadotropin (hCG) test at screening or prior to dosing abbr de ante meridiem (AN ). Agrees to use one of the contraception methods listed by Investigator/designee for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until seven days after the drug administration. or has only same-sex partners, when this is her preferred and usual lifestyle.
* Body mass index (BMI) between 18-27.0 kilogram per meter (kg/m^2) according to Quetelet.
* Volunteers should be healthy as determined by their medical evaluation done by the physicians in the center and by their safety labs results done at a certified local laboratory.
* Variation limits within normal ranges on their screening visit are: Blood pressure (BP) (seating) between 90 and 130 millimeters of mercury (mm Hg) for Systolic pressure and between 60 and 90 mmHg diastolic pressure, heart rate (HR) between 55 and 100 beats per minute (bpm) and respiratory rate (RR) between 14 and 20 per minute.
* Safety laboratory tests to be done include: Hematology: Complete blood count with differential, Hemoglobin, Hematocrit, platelet count, etc; Blood chemistry: Albumin, Alkaline phosphatase, aspartate-aminotransferase (AST), alanine aminotransferase (ALT), Urea, Calcium, Chloride, Glucose, Phosphate, Potassium, Serum creatinine, Sodium, Total bilirubin, Total protein, etc; Urinalysis: pH, Specific gravity, Protein, Glucose, Ketones, Bilirubin, Occult blood and cells, Nitrite, Urobilinogen, Leukocytes, Microscopic examination; Hepatitis B and C tests; human Immunodeficiency Virus (HIV) test; Serum pregnancy test; Drug abuse test; Alcohol detection test; Urine Pregnancy test; ECG; Chest X ray. Normal variation limits for laboratory values will be +/- 10% from normal range, unless the principal investigator (PI) considers another deviation as clinically non-significant. In that case, values should be documented in the volunteer's clinical file as well as the decision to include the subject prior consult with GlaxoSmithKline (GSK) Medical Monitor. For safety reasons and as per the PI criteria additional ECG or safety labs may be performed.

Exclusion Criteria:

* Subjects with changes on their vital signs compared to what obtained in the screening visit.
* Volunteers that not comply with all the inclusion criteria described previously
* Volunteers with history of clinically relevant cardiovascular, renal, hepatic, muscular, metabolic. Clinically relevant hematologic, gastrointestinal, neurological, endocrine, pulmonary, mental disease or any other organical abnormality. Volunteers with muscular traumatism within 21 days before the study.
* Volunteers that require any drug during the study, besides the study drug.
* Volunteers with dyspepsia, gastritis, esofagitis, duodenal o gastric ulcers.
* Volunteers that have received hepatic metabolism drug inhibitors or inducers within 30 days of the beginning of the study and that have received drugs that may alter urinary pH, like antiacids with sodium bicarbonate, potasium citrate and certain diuretics
* Volunteers who received any drug and that 7 half lives have not been completed at the beginning of the study.
* Volunteers who have ALT, alkaline phosphatase and bilirubin <= 1.5x upper limit of normal range (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Corrected QT interval duration (QTc) values of triplicate ECGs obtained over a brief recording period: QTc < 450 milliseconds (msec); or QTc < 480 msec in subjects with Bundle Branch Block.
* Volunteers that might have required to be hospitalized for any reason within 6 months before the beginning of the study
* Subjects with a previous participation in another research study within 60 days prior to the beginning of the study.
* Subjects allergic to any food, drug and/or substance
* Subjects with known history of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects who consume alcohol, coffee, grapefruit, nicotine, orange or metilxantines containing substances (coffee, tea, chocolate, cola products, broiled products etc) within 72 hours prior to their confinement period and until the end of the study.
* Subjects that might have lost or donated 450 ml of blood within the 60 days prior to the beginning of the study.
* Alcohol or drug abuse history
* Volunteers who require special meals (vegetarian).
* Unwillingness or unable to understand the nature, objectives of possible consequences of the study.
* Evidence of not being able to cooperate during the study
* Positive alcohol, drug abuse and/or pregnancy tests
* Breast feeding
* Volunteers under any kind of hormonal therapy
* Volunteers not registered at COFEPRIS web page

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2014-09-08 (Actual); Study Completion 2014-09-08 (Actual)

PRIMARY OUTCOMES:
Composite of PK parameters for eltrombopag | Serum Pharmacokinetic (PK) samples will be collected pre-dose and then samples will be obtained 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 8.0, 12, 16, 24, 48, 72 and 96 hours after drug administration
  Following PK parameters will be assessed: Area under the concentration-time curve from time zero to last time of quantifiable concentration within a subject (AUC[0-t]), area under the curve (concentration/time) from time 0 extrapolated to infinity (AUC[0 inf]), maximum observed concentration (Cmax) and time to Cmax (tmax)

SECONDARY OUTCOMES:
Incidence and nature of adverse events (AEs) and Serious adverse events (SAEs) | Up to Day 12
  AEs and SAEs will be collected from the screening until the follow-up visit
Monitoring vital signs | Up to Day 12
  Vital signs assessments included temperature, systolic and diastolic blood pressure, and pulse rate measurements
Electrocardiograms (ECG) assessments | Up to Day 12
  Single 12-lead ECGs will be obtained over a brief (eg, 5-10 minute) recording period at each study visit.
Clinical laboratory parameters | Up to Day 12
  Clinical laboratory parameters will include hematology, clinical chemistry and urine analysis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mexico City, Mexico

REFERENCES:
- See also: Results for study 200338 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200338?search=study&search_terms=200338#rs